CLINICAL TRIAL: NCT03695263
Title: Massive Individualized N-of-1 Experiments Using HackYourHealth: A New Paradigm for Promoting Health and Well-Being
Brief Title: Massive Individualized N-of-1 Experiments (MINEs)
Acronym: MINEs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of California, San Francisco (Other); University of California, San Diego (Other); Brown University (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1255435
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Stress, Psychological; Happiness; Cognition
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Each participant will enroll in a personalized ("N-of-1") crossover trial.
Masking Description: The analysis will proceed automatically without knowledge of which 3-day treatment periods were associated with one of the five interventions and which were associated with the subject's usual activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N-of-1 Trial (Experimental): Multiple crossovers between one of the available intervention options (mindfulness meditation, gratitude journaling, physical activity, laughter therapy, or random acts of kindness) and usual activities
  Interventions: Behavioral: Choice of one of five behavioral interventions

INTERVENTIONS:
Behavioral: Choice of one of five behavioral interventions — All participants will choose one of the five intervention options.

SUMMARY:
The project will enroll up to 10,000 adult volunteers in individualized experiments (N-of-1 trials) designed to assess the individual-level effects of any of five interventions on three outcomes. The five interventions are: gratitude journaling, mindfulness meditation, random acts of kindness, physical activity, and laughter therapy. The three outcomes are stress, cognitive focus, and happiness. Each participant will engage in the selected activity in 3 day intervals, separated at random by 3 day intervals of usual activity, for a total of six 3-day periods (18 days).

DETAILED DESCRIPTION:
N-of-1 trials (single patient crossover experiments) are a uniquely powerful technique for estimating treatment effects in the individual. N-of-1 trials have been offered to hundreds or perhaps thousands of patients worldwide, but never at scale. HackYourHealth is a tool that supports the conduct of simple N-of-1 self-experiments to test if healthy activities that work in general (i.e., mindfulness meditation, physical activity, gratitude journaling, random acts of kindness, and laughter therapy), improve psychological well-being (stress, focus, happiness) in specific individuals. The tool supplies the experimental design, facilitates data analysis, and channels feedback to participants. The tool is flexible enough to support Massive Individualized N-of-1 Experiments (MINEs) at scale. Working with WNYC Radio in New York City, we will recruit and run 18-day N-of-1 trials up to 10,000 individuals. The purpose of this study is to conduct a formative evaluation of HackYourHealth in terms of its perceived usefulness and to explore heterogeneity in intervention response across the sample. We anticipate that the results will: 1) identify useful behavioral interventions for individual participants; 2) help to estimate generalizable treatment effects for the interventions of interest; 3) assess heterogeneity of treatment effects across subgroups; and 4) elucidate the user experience with N-of-1 trials. When complete, the study will support additional proposals designed to assess the utility of MINEs as applied to additional conditions and treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Living anywhere in the United States
* Using a smartphone
* Having regular access to internet on their phone
* Able to read and write in English

Exclusion Criteria:

There are no exclusion criteria, except that patients with pre-existing cardiovascular disease will be cautioned not to engage in new types of physical activity without consulting a physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Stress | 18 days
  How stressed are you feeling today? (single item Likert scale).Stress will be measured using a single Likert-type question that ranges from 0-10, For stress 0 (not at all) represents a better outcome and 10 (as much as possible) represents a worse outcome.
Focus | 18 days
  How focused are you feeling today? (single item Likert scale).Focus will be measured using a single Likert-type question that ranges from 0-10. For focus 0 (not at all) represents a worse outcome and 10 (as much as possible) represents a better outcome.
Happiness | 18 days
  How happy are you feeling today? (single item Likert scale).Happiness will be measured using a single Likert-type question that ranges from 0-10. For happiness 0 (not at all) represents a worse outcome and 10 (as much as possible) represents a better outcome.

SECONDARY OUTCOMES:
User burden | Within 1 to 28 days of N-of-1 trial completion
  User Burden Scale (UBS) - The UBS is a 20-item scale, with 6 individual sub-scales, that assesses the burden placed on users by computing systems. The 6 burden-related constructs evaluated through the sub-scales are: (1) difficulty of use (2) physical (3) time and social (4) mental and emotional (5) privacy (6) financial The UBS uses two 5-point scales ranging from 0-4 (Never - All of the time; Not at all - Extremely). Total score is a sum of responses to all questions in the scale. A higher score indicates a higher level of user burden. The maximum score is 80 and minimum is 0.
  User burden can be explored by sub-scales to explore which construct is contributing most to user burden. In such a case, scores for each sub-scale are computed by calculating the mean for items within each sub-scale.

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Kravitz, MD, MSPH, Principal Investigator — UC Davis Division of General Medicine
Locations (1):
- UC Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No